CLINICAL TRIAL: NCT05765942
Title: Expression of microRNAs (146a and 155) and Cytokines in the Tissue Surrounding Dental Implants Diagnosed With Peri-implantitis
Brief Title: MicroRNAs and Cytokines in Peri-Implantitis Tissue
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, munir nasr, Principal Investigator, University of Baghdad
Other Study IDs: 534622
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Implant surgery for harvesting healthy implant tissue (group HP): the preoperative mucosal thickness will be measured clinically using a periodontal probe. A crestal incision will be performed, and a full-thickness flap will be elevated. Following the osteotomy, one or more implants measuring 4.5 or 5.0 mm in diameter will be placed. The implant platform will be positioned 0.5 mm below the bone level. A narrow-diameter healing abutment designed specifically for this study will be screwed in at 20 N, and flaps will be repositioned and sutured to obtain optimal adaptation of the mucosa to the titanium abutment. Healthy tissue samples will be harvested after 2 months of healing. Before the surgery, a guide pin will be connected to each healing abutment, attached to a circular punch 5 mm wide and with a cutting edge, which screwed apically around the abutment. Hence, a 1.5 mm thick collar of peri-implant soft tissue will be harvested Then, a new 4.5-5.0 mm-wide smooth-surfaced healing abutment will be connected to the implant directly.
- Implant surgery for harvesting peri-implantitis tissue (group PP): In each patient, at least one implant site demonstrating signs of peri-implantitis will be selected for biopsy. The site will be anesthetized and two parallel incisions, about 3mm apart, will be made with a 15C scalpel blade through the soft tissue until bone contact would be achieved. The 2 incisions will be connected with a perpendicular incision that will be placed at a distance of 4 mm from the proximal surface of the implant. The biopsies, including the entire supra-crestal soft tissue portion of the diseased site, will be carefully retrieved

SUMMARY:
Peri-implantitis is a non-linear and accelerating pattern of loss of supporting bone tissue associated with clinical signs of inflammation and increased probing depths compared to baseline measurements. It can present as an asymptomatic condition with infection and fast progression of bone resorption or clinically symptomatic with mucosal inflammation, redness, edema, mucosal enlargement, bleeding on probing (BOP), suppuration, increased probing depth, and radiographic bone loss. The host immune defense against bacterial challenge is responsible for the damage, and the local immune-inflammatory process is associated with disrupted bone remodeling. New studies looking for predictive and accurate early biomarkers for this pathology have the utmost relevance. David Baltimore et al. proposed a feedback loop involving miRNA-146a and TLR signaling, which has been shown to be up-regulated in inflammatory diseases such as osteoarthritis and rheumatoid arthritis.

miRNA-146a and miRNA-155 were the first miRNAs identified to be induced in immune cells stimulated by TLRs and proinflammatory cytokines. Precision medicine uses molecular research and different biomarkers, population studies, and big data analysis to recreate complex disease models. Several studies have compared the miRNA profiles of patients with periodontitis with healthy patients. Although periodontitis and peri-implantitis share many features, researchers' findings of periodontitis are not necessarily applicable to peri-implantitis. In fact, based on emerging evidence, peri-implantitis, and periodontitis exhibit several key differences, including their histopathological and molecular characteristics. Considering the aforementioned analysis, inflammatory miRNAs may be differentially expressed in peri-implantitis tissue compared with healthy gingival tissue. This study will investigate the gene expression levels of miRNA-146a and miRNA-155 and their correlation with inflammatory levels of their target genes in human gingival tissue surrounding dental implants diagnosed with peri-implantitis and health.

DETAILED DESCRIPTION:
MiRNAs are small non-coding RNA molecules that are approximately 18-22 non-transcribed spacer NTS long. These single-stranded molecules regulate gene expression by binding to the complementary sequences in the 3-untranslated or coding region of the target mRNAs, leading to either blockade of translation or induction of target mRNA degradation. Therefore, miRNAs participate in not only physiological processes within cells and tissues but also pathological processes. According to previous reports, miRNAs are specifically involved in many inflammatory and bone-related diseases, such as rheumatoid arthritis, osteoporosis, and periodontitis.

The miRNA-146 family is composed of two members, miRNA-146a and miRNA-146b that are located on chromosomes 5 and 10, respectively. proposed a feedback loop involving miRNA-146a and TLR signaling. They found the induction of transcription of miRNA-146a by lipopolysaccharide LPS, tumor necrosis factor-alpha (TNFa) and interleukin-1b (IL-1b) is dependent on NF-kb, and that in turn, miRNA-146a potentially targets tumor necrosis factor receptor-associated family (TRAF6) and interleukin-1 receptor-associated kinase (IRAK1), implicating it as a negative regulator ﬁne-tuning the immune response. As stated, too strong or too prolonged induction of the innate immune response can have detrimental effects resulting in acute and chronic inﬂammatory disorders. The high expression of miRNA-146a is up-regulated in many inﬂammatory diseases such as osteoarthritis and rheumatoid arthritis (RA), the latter involving up-regulation following stimulation with inﬂammatory cytokines such as TNF-a and IL1-b. Interestingly, a polymorphism in the 3-untranslated region (3-UTR) of the mRNA encoding the miR-146a target IRAK1 is associated with susceptibility to Rheumatoid Arthritis and psoriatic arthritis.

MiRNA-146a and miRNA-155 were the ﬁrst miRNAs identiﬁed to be induced in immune cells stimulated by TLRs and proinﬂammatory cytokines. In human and murine immune cells, miRNA-155 can be classiﬁed as an early response gene, since its expression is highly induced within 2 h of TLR activation (TLR2, TLR3, TLR4, and TLR9). MiRNA-155 negatively regulates TLR-signaling by targeting key signaling molecules, including TAB2, MyD88, and NF-kb subunit p65. Overexpression of miRNA-155 suppresses the production of the proinﬂammatory cytokines IL-8 and TNF-a, whereas IL-10, which exerts anti-inﬂammatory properties, inhibits miR-155 expression to maintain homeostasis. MiR-155 also facilitates CXCL12 signaling through the inhibition of SHIP-1, a negative regulator of TLR-induced signals. Moreover, SHIP-1 regulation by miR-155 controls the pathogenesis of experimental colitis, suggesting that miR-155 can also have proinﬂammatory functions.

The advances made in proteomics, genomics, and molecular biology aid in the control and treatment of the disease by taking advantage of precision or stratified medicine, i.e. "segregating the individuals into subpopulations who vary in their disease susceptibility and response to a precise treatment". Precision medicine uses molecular research and different biomarkers, population studies, and big data analysis to recreate complex disease models. It seems reasonable to expect that in the future, the accuracy, predictive values, and advantages of these predictive models which include new molecular candidates could benefit and improve the control of different multifactorial and complex diseases, such as peri-implantitis. Indeed, this approach has been considerably developed in oncology and genetic diseases, but it is still under progress in the dental field. Expanding the research of new molecules and biomarkers in peri-implant tissues would allow us to monitor the clinical status of the implants, to classify them as well as the patients according to their real risk of developing biological complications. In this regard, an important class of gene modulators that have been scarcely explored in the context of periimplantitis include miRNAs.

Several studies have compared the miRNA profiles of patients with periodontitis with healthy patients. Although periodontitis and peri-implantitis share many features, researchers' findings of periodontitis are not necessarily applicable to peri-implantitis. Based on emerging evidence, peri-implantitis, and periodontitis exhibit several key differences, including their histopathological and molecular characteristics. Considering the aforementioned analysis, inflammatory miRNAs may be differentially expressed in peri-implantitis tissue compared with healthy gingival tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Peri-implant health (control group):

   * Adult patient age between >18years.
   * Having one or more missing teeth will be replaced with dental implants.
   * Having adequate bone quality and availably for implant placement of 4.5-5 mm diameter and 8.5-13 mm length.
   * Having keratinized mucosa of at least 3mm.
   * Having no systemic disorders contraindicating to have peri-implant therapy.
2. Peri-implantitis (test group):

   * Adult patient age between >18 years old.
   * Having at least one implant with > 1 year in function.
   * Presence of bleeding and/or suppuration on gentle probing.
   * Increased probing pocket depth (PPD) compared with previous baseline data
   * Presence of bone loss beyond initial bone remodeling levels.

In the absence of previous examination data diagnosis of peri-implantitis can be based on the combination of:

* Presence of bleeding and/or suppuration on gentle probing.
* PPD of ≥6 mm.
* Bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant.

Exclusion Criteria:

* Chronic inflammatory diseases such as : type 1 or 2 diabetes, cardiovascular or autoimmune diseases, and active infectious diseases.
* Systemic or topical antimicrobial/anti-inflammatory therapy for the 3 months prior to the beginning of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients will be selected from private clinics in Baghdad, seeking dental implant treatments. The peri-implant healthy group (control group) will involve those who are seeking to replace missing teeth with dental implants. While, the peri-implantitis patients (test group) will involve those who will be diagnosed with peri-implantitis and need surgical intervention during their follow up visits.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of miRNAs expressed in gingival tissue | 4 days
  Level of miRNA (146a-5p and 155-5p) per fold change expressed in gingival tissue surrounding dental implants diagnosed with peri-implantitis and health.

SECONDARY OUTCOMES:
Level of mRNAs expressed in gingival tissueLevel | 4 days
  Level of mRNA (TLR-4, IL-1b, TNFa and IL-10) per fold change expressed in gingival tissue surrounding dental implants diagnosed with peri-implantitis and health.

CONTACTS AND LOCATIONS:
Locations (1):
- Munir, Baghdad, Iraq